CLINICAL TRIAL: NCT02552342
Title: Efficacy of Methylprednisolone in Severe Community-acquired Pneumonia，A Multi-center Randomized Controlled Trial
Brief Title: Corticosteroid Therapy for Severe Community-Acquired Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Tianjin Medical University General Hospital (Other); Cangzhou Central Hospital (Other); Cangzhou People's Hospital (Other); Affiliated Hospital of Hebei University (Other); Nantong University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Northern Jiangsu People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); Taishan Medical University Affiliated Hospital (Other); Tianjin Third Central Hospital (Other); Jinhua Central Hospital (Other); Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-836
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone (Active Comparator): This group was entitled to receive methylprednisolone 80mg/day for 3 days，then 40mg/day for 3 days
  Interventions: Drug: methylprednisolone
- Placebo (Placebo Comparator): This group was meant to receive placebo (sterile normal saline in a volume equal to the study drug
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: methylprednisolone
  Other Names: Solu-Medrol
  Arms: methylprednisolone
Drug: Normal saline
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of the present study is to assess the efficacy of methylprednisolone as an adjuvant therapy in patients with severe community-acquired pneumonia (CAP) (PSI 4-5).

The hypothesis of the study is that methylprednisolone can decrease the mortality of severe CAP without any significant side effects,with reduction of the time to clinical stability and failure rate of treatment.

ELIGIBILITY:
Inclusion Criteria:

* community-acquired pneumonia
* PSI score：4-5
* with at least one of following conditions：①CRP ≥150 mg/L,②oxygen index ≤250 , ③bilateral or multi-lober infiltrates in chest image,④ area of pulmonary infiltrates increase >50% with 48 hous,⑤fever higher than 39℃ exceed 72 hours

Exclusion Criteria:

* nosocomial Pneumonia
* aspiration pneumonia
* acute burn injury
* gastrointestinal bleeding within the past three months
* uncontrolled diabetes mellitus
* pregnant or breast feeding
* a condition requiring treatment with greater than 0.5 mg/kg/d of prednison or its equivalent
* severe immunosuppression (human immunodeficiency virus infection, immunosuppressive conditions or medications)
* active tuberculosis
* preexisting medical condition with a life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhong Yu, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China